CLINICAL TRIAL: NCT06022120
Title: Health Literacy Among Youth (Danish: Sundhedskompetencer Blandt Unge)
Brief Title: Health Literacy Among Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holbaek Sygehus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: REG-068-2023
Record Dates: First submitted 2023-08-09; First posted 2023-09-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Health Knowledge, Attitudes, Practice; Health Behavior; Health Literacy; Health-Related Behavior
Keywords: Health Literacy; Health behavior; Intervention; School context; Youth
MeSH Terms: conditions — Behavior; Health Behavior

STUDY DESIGN:
Intervention Model Description: Using a stepped-wedge design, participants at the enrolled schools function as their own control. Thus, the effect of the intervention is evaluated as in an RCT design. All participants are asked to indicate whether they want to participate in the scientific evaluation of the intervention. Those who wish to participate are invited to the data collection containing: Signing of consent and answering questionnaires. No preparation is required of the participants before data collection begins. Smaller groups of students and teachers participate in focus groups as part of the process evaluation. All intervention activities take place at the participants' school. Calculation, analysis and interpretation of data will take place at the Department of Occupational and Social Medicine, Holbæk Hospital.
  The intervention activities are developed by a student commitee, accoording to a participatory approach and following the Work Health Improvements Network concept.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- An integrated health literacy intervention (Other): Intervention: A group of students at each school will develop and implement their own project activities at meetings two times during the intervention. Activities are implemented in schools for all students.
  Interventions: Behavioral: An integrated health literacy intervention
- Reference (No Intervention): No intervention activities

INTERVENTIONS:
Behavioral: An integrated health literacy intervention — The intervention investigates the effect of the Australian WorkHealth Improvement Network (WIN) program and the Total Worker Health (TWH) concepts in a Danish contexts among students at risk of poorer health outcomes compared to their peers with stronger literacy skills.
  Arms: An integrated health literacy intervention

SUMMARY:
The linkage between lower educational levels and poorer health has been highlighted as a mechanism contributing to social inequality in health. However, more research on this mechanism among youth is needed, e.g. to ensure timing of primary prevention of diseases. Additionally, health literacy (HL) has been increasingly recognized as a means of reducing health inequalities. However, knowledge on best practice for HL interventions among youth is scarce. The aim of this project is to develop, test, and evaluate an integrated, participatory intervention to improve HL among young adults in Danish school settings.

DETAILED DESCRIPTION:
OBJECTIVE This project aims to develop, test, and evaluate an integrated, participatory intervention to improve health literacy (HL) through health promoting activities among young Danes in school settings.

Research questions:

* What are the HL needs of young adults in Danish FGU or similar school settings?
* Is an integrated, participatory intervention approach feasible in FGU schools or similar settings and effective to improve the HL of the students?

BACKGROUND Social inequality in health refers to health differences between social groups, and the pattern in which those from economically and socially poorer backgrounds run higher risks of premature death and illness. Furthermore, the strong linkage between lower educational levels and poorer health has been highlighted as one of the mechanisms contributing to social inequality in health. In 2018, approximately 50,000 Danes aged 15-24 years were Not in Employment, Education or Training (NEET) and almost 20% of all Danish 25-year olds had not completed a secondary education. Thus, a relatively large proportion of Danish youth were at risk of exclusion from the labour market, lower income, and thereby also reduced health.

To support young adults who are NEET, preparatory basic educational institutions (Danish: Forberedende grunduddannelse (FGU)) were initiated in 2019. One report finds that FGU students are disadvantaged in terms of socio-demographic and educational factors compared to their peers, and 50% of FGU students have special educational needs, including psychiatric diagnoses. Hence, students at FGU educations represent a group of young adults who are at particular risk of adverse health outcomes.

Health Literacy (HL) is now well-established as a modifiable factor that contributes to the maintenance of good health across the life course, and globally, there has been an increasing acknowledgement of HL as a means of reducing health inequalities. However, HL follows a social gradient, e.g. inadequate HL is more prevalent among vulnerable populations, such as persons with low education. The World Health Organization (WHO) has stated a need for development of national strategies to strengthen HL in all populations and in educational contexts, and more countries have now included HL in national health strategies. However, the Danish health authorities have not shown similar interest in HL, and their focus have primarily been on organizational HL responsiveness and not on the individual's HL. With the increasing calls for more actions on addressing HL and health inequality, school-based HL interventions have emerged. However, such HL interventions have so far faced implementation challenges, and there is a shortage of clarity about which intervention strategies are the most effective in improving HL among children and young adults.

METHODS In this project, an integrated, participatory intervention to improve HL among young Danes at FGU schools or similar contexts is developed, tested and evaluated by use of mixed-methods and the UK Medical Research Counsil's framework for developing and evaluating complex interventions. The integration means that all intervention activities have a preventive and health-promoting element. The intervention concept is developed by The American Total Worker Health (TWH) and the Australian WorkHealth Improvement Network (WIN) program. Recently, the Department of Occupational and Social Medicine (ASMA) at Holbæk Hospital tested the WIN concept in a Danish context among adult employees with little or no education, and preliminary analyses showed promising results. As the intervention concept is very flexible and is based on local adaption, we assume that it is possible to implement in two Danish FGU schools or similar settings.

To this date, one FGU and one technical school has expressed willingness to participate in the intervention.

The intervention involves three phases:

Phase 1: The needs assessment includes: 1) A systematic review about HL interventions among youth in school settings; 2) Individual, semi structured interviews or focus groups with local experts (e.g. teachers at FGU schools), who are strategically selected based on their knowledge about the organizational structure and experience with the target group, to clarify the HL needs from a professional perspective; 3) Two focus groups at each school (in total, n=24-28) with the target group, i.e. students, are conducted pre the intervention to clarify the HL needs of the students. Qualitative data are analyzed in NVivo software by use of thematic network analysis and interpreted by use of social practice theory, which has previously been used to analyze complex relationships between intervention elements (competencies, materials and meanings) and social context in complex interventions.

Phase 2: Program implementation: The intervention is implemented after adjustment according to the needs assessment. The integrated intervention design allows for local adaption, i.e. the specific focus point for the intervention activities will be based on issues in the local context brought up by the participants themselves. Additionally, the intervention concept follows a systematic, participatory approach where participants are supported to develop their own HL initiatives. The intervention activities includes:

1. Establishment of a HL committee: A group of students (6-7) and a teacher join a HL committee at each school. The HL committee participate in two 3-hours workshops where they will be educated and trained in collaborative methodology and WIN concepts (particularly in the first workshop).
2. Development of own initiatives: During the workshops, the HL committee will develop own initiatives to improve HL among all students at each school.
3. Implementation of initiatives: Between the workshops, the HL committee will test and implement their initiatives, e.g. using the Model of Improvement and the plan-do-study-act (PDSA) cycle (as described below). In every implementation period, the HL Committee at each school meets and discuss the implementation. The students in the HL committee will document changes and barriers and facilitators to the implementation by taking photos and do an on-going evaluation.

The Model of Improvement consists of a brainstorming part including three key questions aiming to guide the assessment of which initiatives to focus on: 1) What are we trying to accomplish?, 2) How will we know that a change will lead to an improvement?, and 3) What changes can we make that will result in an improvement?). The second part is the "test part", which consist of the PDSA cycles: 1) Plan: Thorough planning of the initiative, clarification of expectations of outcomes, and agreements on data collection, 2) Do: Implementation of the planned actions as well as data collection, 3) Study: Reflection on effect and learning, data analysis, and identification of unintended negative and positive consequences, and 4) Act: Assessment of either continuation of implementation, adjustments, or testing a new initiative. The experiences from each cycle will systematically be transferred to the next. Thus, continuous improvements and/or adjustments will be conducted.

Phase 3: Process- and effect evaluation: Pre-, during (x2), and post the intervention, questionnaire data are collected among all students at the schools. Until baseline, participants function as their own controls as in a RCT design. Questionnaire data are analyzed in linear mixed models that take into account repeated measurements as well as inter- and intra-effect differences among the participants. Focus groups with 6 students at each school are conducted to evaluate the implementation of the intervention and its feasibility by use of a realist evaluation approach.

ELIGIBILITY:
Inclusion Criteria:

* Providing an informed signed consent prior to participation.
* Student at one of the enrolled schools
* 15-25 years of age or turns 15 during the project period.

Exclusion Criteria:

* Under the age of 15 and does not turn 15 during the project period.
* above the age of 25 before the project period starts.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 176 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Health Literacy | Data on health literacy are collected at baseline and follow up data are collected 3 and 6 months after randomization.
  Change of health literacy level measured by HLS19-Q12 (Danish version), ranging from 1-4, with higher scores indicating a higher level of health literacy, from baseline to 3 and 6 months after randomization.

SECONDARY OUTCOMES:
Self-perceived health | Data on self-perceived health are collected at baseline and follow up data are collected 3 and 6 months after randomization.
  In a questionnaire participants are asked: "All in all, how do you think your health is?". Change of self-perceived health (SF-36, Danish version, by Bjørner et al. 1997), ranging from 0-5 with a higher scores indicating a worse health outcome, from baseline to 3 and 6 months after randomization.
Life satisfaction | Data on life satisfaction are collected at baseline and follow up data are collected 3 and 6 months after randomization.
  In a questionnaire participants are asked: "How satisfied are you with your life?". Change of life satisfaction, ranging from 0-10, with higher numbers indicating a higher life satisfaction, from baseline to 3 and 6 months after randomization.
Mental health | Data on mental health are collected at baseline and follow up data are collected 3 and 6 months after randomization.
  In a questionnaire participants are asked to indicate their mental health by answereing to what degree they agree with four statements: 1) I was happy last week, 2) I felt my friends were not freindly and did not want to spend time with me, 3) I felt sad, 4) It was not easy to get started this week. Change of mental health, ranging from 1-4, with higher numbers indicating worse mental health, from baseline to 3 and 6 months after randomization.
Self efficacy | Data on self efficacy are collected at baseline and follow up data are collected 3 and 6 months after randomization.
  In a questionnaire participants are asked to indicate to what degree they agree with three statements: 1) Your are good at solve unexpected problems, 2) You can solve most problems, if you really want to, 3) despite what happens in your life, you feel like you will be able to solve it. Change of self efficacy, ranging from 1-5, with higher numbers indicating worse outcome, from baseline to 3 and 6 months after randomization.
Ressources for health promotion | Data on ressources for health promotion are collected at baseline and follow up data are collected 3 and 6 months after randomization.
  In a questionnaire, participants are asked about access to healthy food and physical activity facilities. Change in ressources for health promotion, ranging from 1-4, with higher numbers indicating better outcome, from baseline to 3 and 6 months after randomization.
Leisure time physical activity | Data on leisure time physical activity are collected at baseline and follow up data are collected 3 and 6 months after randomization.
  In a questionnaire, participants are asked about their level of physical activity in leisure time. Change in leisure time physical activity, ranging from 1-6, with higher numbers indicating a better outcome, from baseline to 3 and 6 months after randomization.
Alcohol consumption | Data on alcohol consumption are collected at baseline and follow up data are collected 3 and 6 months after randomization.
  In a questionnaire, participants are asked about their alcohol consumption. Change in alcohol consumption ranging from 1-7, with higher numbers indicating a worse outcome, from baseline to 3 and 6 months after randomization.
Nicotine and weed consumption | Data on nicotine/weed consumption are collected at baseline and follow up data are collected 3 and 6 months after randomization.
  In a questionnaire, participants are asked about their nicotine and weed consumption. Change in nicotine/weed consumption ranging from 1-4, with higher numbers indicating a worse outcome, from baseline to 3 and 6 months after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian Rueskov Poulsen, Principal Investigator — Holbæk Sygehus
Locations (1):
- Department of Occupational and Social Medicine, Holbaek Hospital, Holbæk, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No
We do not plan to share any individual participant data with other researchers.